CLINICAL TRIAL: NCT06230952
Title: Reliability of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Bath Ankylosing Spondylitis Functional Index (BASFI) Applied by Tele-Assessment Method in Patients With Axial Spondyloarthritis
Brief Title: Reliability of BASDAI and BASFI Applied by Tele-Assessment Method in Axial SpA Spondyloarthritis
Status: Completed | Type: Observational
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Yasemin ACAR, Research assistant, Siirt University
Other Study IDs: 2023/39-19
Record Dates: First submitted 2024-01-16; First posted 2024-01-30 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; BASDAI; BASFI; self assessment; tele-assessment; reliability
MeSH Terms: conditions — Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- axial spondyloarthritis patients: patients diagnosed with axial spondyloarthritis
  Interventions: Other: BASDAI and BASFI reliability

INTERVENTIONS:
Other: BASDAI and BASFI reliability — The study will be carried out on volunteer patients who are diagnosed with axial spondyloarthritis and are followed up in the outpatient clinic of Dokuz Eylül University, Department of Internal Medicine, Rheumatology and Immunology Department, and who meet the inclusion criteria. Patients who volunteer to participate in the study will be contacted by phone and BASDAI and BASFI questionaires will be administered.

SUMMARY:
The goal of this observational study is to investigate the reliability of BASDAI and BASFI questionnaires applied via tele-assessment in axial spondyloarthritis patients.

DETAILED DESCRIPTION:
Telehealth is the provision of healthcare services and clinical practices remotely through information and communication technologies. In recent years, the use of telehealth applications has increased worldwide. Telehealth is an umbrella term that covers practices such as telemedicine, telerehabilitation, and tele-assessment. Tele-assessment has gained importance in terms of monitoring patients with chronic diseases. Although BASDAI and BASFI have been shown to be valid and reliable in AS patients, there is no study in the literature examining the reliability of BASDAI and BASFI applied via tele-assessment. The aim of our study is to investigate the reliability of BASDAI and BASFI questionnaires administered via tele-assessment in axial SpA patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Axial spondyloarthritis according to the Assessment in SpondyloArthritis international Society (ASAS) criteria
* Volunteering to participate in the study
* Being between the ages of 20-60

Exclusion Criteria:

* Having another systemic, orthopedic, neurological or cognitive disease other than axial spondyloarthritis
* Pregnancy
* The patient wishes to withdraw from the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: It was planned to include at least 100 axial SpA patients in the study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline and after 24 hours after baseline assessment
  Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a reliable and sensitive index developed to evaluate the activity and progression of the disease. The BASDAI is a 6-item composite index that measures fatigue, neck, back, hip pain, peripheral joint pain/swelling, and morning stifness. The final BASDAI score ranges from 0 to 10, and higher scores represent higher disease activity.
Bath Ankylosing Spondylitis Functional Index (BASFI) | Baseline and after 24 hours after baseline assessment
  BASFI is an easy-to-apply, sensitive and reliable self-report questionnaire developed to evaluate physical function in AS patients. It consists of a total of 10 items, eight assessing functionality and two assessing the patient's ability to cope with daily life. The BASFI Score is the avarage of the 10 items and ranges between 0 and 10, with higher scores indicating greater functional limitation.

SECONDARY OUTCOMES:
Age | Baseline
  Age in years
Disease duration | Baseline
  Disease duration in years
Medications | Baseline
  The medications used by patients will be recorded
weight | Baseline
  weight (kg)
height | Baseline
  height (m)
Education | Baseline
  Education level of patients will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ACAR, PhD, Study Director — Siirt University
Locations (1):
- Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acar Y, Ilcin N, Sari I. Reliability of the Bath Ankylosing Spondylitis Disease Activity Index and the Bath Ankylosing Spondylitis Functional Index administered via tele-assessment in patients with axial spondyloarthritis. Physiother Theory Pract. 2025 Dec;41(12):2585-2594. doi: 10.1080/09593985.2025.2536319. Epub 2025 Jul 21. PMID 40686331